CLINICAL TRIAL: NCT02087228
Title: Evaluation of the Endometrial Cavity After Endometrial Ablation
Acronym: Postablation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor and Principle Investigator mutually agreed to terminate study and patients are no longer examined/treated
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 013-053; BRI-2013-1979 (Other: Baylor Research Institute)
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Menorrhagia
Keywords: Endometrial ablation, menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrothermal ablation (Experimental): Uterine ablation performed with a device that circulates heated water inside the uterus
  Interventions: Device: Genesys HydroTherm Ablator
- radiofrequency energy (Active Comparator): ablation performed with a device that uses radiofrequency energy.
  Interventions: Device: radiofrequency energy ablation device

INTERVENTIONS:
Device: Genesys HydroTherm Ablator — Heated water is circulated inside the uterus to destroy the lining of the uterus
  Arms: Hydrothermal ablation
Device: radiofrequency energy ablation device
  Arms: radiofrequency energy

SUMMARY:
The purpose of this study is to evaluate the shape, size and appearance of the inside of the uterus six months following an endometrial ablation procedure. Half of the participants will have their ablation performed with a hydrothermal ablation device and the other half will have their ablation performed with a device that uses radiofrequency energy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the shape, size and appearance of the inside of the uterus six months following an endometrial ablation procedure. Half of the participants will have their ablation performed with a hydrothermal ablation device and the other half will have their ablation performed with a device that uses radiofrequency energy. Participants are randomly assigned to one or the other device.

A vaginal ultrasound will be performed before the procedure and again at six months post-procedure.

The inside of the uterus will be visualized via hysteroscopy before the procedure and again at six months post-procedure. Measurements will be taken and the investigator will compare photos taken pre-procedure and six months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women Not pregnant and no future pregnancy desired Willing to randomize the device used for the ablation Willing to undergo diagnostic hysteroscopy with office-based anesthesia 6 months post-ablation

Exclusion Criteria:

* Pregnancy or desiring future pregnancy Endometrial hyperplasia Presence of active endometriosis Active pelvic inflammatory disease Previous endometrial ablation procedure

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Visualization of the inside of the uterus | 6 months post-ablation
  The inside of the uterus will be visualized via hysteroscopy to determine the amount of scarring

SECONDARY OUTCOMES:
Measurments of endometrial thickness | 6 months post-ablation
  Measurements will be taken of the uterine cavity length and endometrial thickness

CONTACTS AND LOCATIONS:
Overall Officials: Delbert A Johns, M.D., Principal Investigator — Texas Health Care, Baylor Research Institute
Locations (1):
- Texas Health Care, Fort Worth, Texas, United States